CLINICAL TRIAL: NCT05275322
Title: Online Group Psychological Intervention for People With Emotional Disorders Using the Unified Protocol
Brief Title: Online Group Psychological Intervention for People With Emotional Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Buenos Aires (Other)
Responsible Party: Principal Investigator, Cristian Javier Garay, Professor, University of Buenos Aires
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDE2120.21
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: To Assess the Clinical Usefulness and Acceptability Level of the UP Online Group Format in Argentina as Well as Participants' Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental)
  Interventions: Behavioral: Unified Protocol
- Waiting list group (No Intervention)

INTERVENTIONS:
Behavioral: Unified Protocol — The Unified Protocol for transdiagnostic treatment of EDs (hereinafter UP) is a transdiagnostic treatment based on emotional regulation published in 2011 by David H. Barlow et al. (Barlow et al., 2011). It consists of eight treatment modules, with five of them being central (mindfulness, cognitive flexibility, countering emotional behaviors, tolerating physical sensations, and emotional exposure).
  Arms: Treatment group

SUMMARY:
Participants will receive an online synchronous group therapy based on the Unified Protocol (UP) model for 11 subsequent weeks, with 90-minute meetings. After every session, they will be sent the chapter with the notions addressed in the session from the UP's patient manual (Barlow et al., 2011) and the scales to work with during the week.

Participants in the waiting list will complete the evaluation scales at the same time as people in the intervention group (before the intervention, in the middle, after the intervention, three months after and six months after). After this period they will receive the group therapy based on the UP.

The group admission criteria are: 1) being 18 years old or older; 2) submitting the informed consent; 3) agreeing to participate in all the scheduled sessions; 4) agreeing to have the sessions recorded (both audio and video) for oversight purposes; 5) submitting a primary diagnosis of an anxiety disorder (e.g., panic disorder; agoraphobia; social anxiety disorder; generalized anxiety disorder; unspecific anxiety disorder), unipolar depression (major depressive disorder; dysthymia), obsessive-compulsive disorder, or post-traumatic stress disorder, according to DSM criteria and disrupting individuals' daily life or causing significant discomfort.

The group exclusion criteria are: 1) comorbidity with psychotic disorders, bipolar disorder, eating disorders, borderline personality disorder, or active severe suicidal ideation, and 2) currently receiving pharmacological treatment. All candidates who are not included in the group will be informed of this decision and will be given information on places to seek treatment. Evaluations will be carried out via video calls on the Google Meet platform, using the MINI (Ferrando et al., 2000) and SCID-II (Grilo, Anez & McGlashan, 2003) diagnostic interviews.

ELIGIBILITY:
Inclusion Criteria:

* 1) being 18 years old or older; 2) submitting the informed consent; 3) agreeing to participate in all the scheduled sessions; 4) agreeing to have the sessions recorded (both audio and video) for oversight purposes; 5) submitting a primary diagnosis of an anxiety disorder (e.g., panic disorder; agoraphobia; social anxiety disorder; generalized anxiety disorder; unspecific anxiety disorder), unipolar depression (major depressive disorder; dysthymia), obsessive-compulsive disorder, or post-traumatic stress disorder, according to DSM criteria and disrupting individuals' daily life or causing significant discomfort.

Exclusion Criteria:

* 1) comorbidity with psychotic disorders, bipolar disorder, eating disorders, borderline personality disorder, or active severe suicidal ideation, and 2) currently receiving pharmacological treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory II | 5 weeks
  Beck Depression Inventory II (BDI II; Beck et al, 2006; Argentine adaptation by Brenlla & Rodríguez, 2006). The BDI II is a questionnaire designed to gauge how severe people's depressive symptoms are. It includes 21 items that probe the typical symptoms of a depressive episode. Every item features 4 options, ranging from 0 (not at all) to 3 (severe, nearly unbearable), on a Likert-type scale. It was validated and adapted to Argentina's population, with an adequate internal consistency and a Cronbach alpha coefficient of .88.
Beck Anxiety Inventory | 5 weeks
  Beck Anxiety Inventory (BAI; Beck et al., 1988; Argentine adaptation by Vizioli & Pagano, 2020). The BAI is an inventory designed to measure the severity of anxiety symptoms. It consists of 21 items, each addressing an anxiety symptom. Every item is rated on a Likert scale answer format that goes from 0 (not at all) to 4 (it upset me very much). This instrument was validated and adapted to Argentina's setting, with a Cronbach alpha coefficient of 0.93.

SECONDARY OUTCOMES:
Positive and Negative Affect Schedule | 5 weeks
  Positive and Negative Affect Schedule (PANAS; Thompson, 2007; Argentine adaptation by Moriondo et al., 2012). The PANAS inventory has been designed to measure affect in a dimensional fashion (negative affect and positive affect). The short version designed by Thompson (2007) and adapted to Argentina by Moriondo et al. (2012) has been chosen. This version covers four dimensions: trait positive affect (five items), trait negative affect (five items), state positive affect (five items), and state negative affect (five items). Every item uses a Likert-type scale rating from 1 (slightly or not at all) through 5 (very much or totally). This instrument features a Cronbach alpha coefficient of .73 (Cronbach alpha coefficient of .84 for Negative Affect and .75 for Positive Affect).
Difficulties in Emotion Regulation Scale | 5 weeks
  Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004; Argentine adaptation by Cremades et al., 2021). This scale measures the extent to which people use several Emotional Regulation strategies. The adapted scale includes 30 self-administered items with a Likert-type five-option scale that goes from 1 (hardly ever) to 5 (almost always) and a six-factor structure, including: (1) impulse control difficulties (six items); (2) limited access to emotional regulation strategies (six items); (3) lacking emotional acceptance (six items); (4) interference in goal-oriented behaviors (four items); (5) lacking emotional awareness (three items), and (6) lacking emotional clarity (six items).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Psychology, University of Buenos Aires, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Celleri M, Cremades CF, Etchevers MJ, Garay CJ. Effectiveness of the Unified Protocol for the transdiagnostic treatment of emotional disorders in online and group format in Argentina: study protocol for a randomized controlled trial. Trials. 2023 Oct 19;24(1):678. doi: 10.1186/s13063-023-07428-4. PMID 37858249